CLINICAL TRIAL: NCT05031611
Title: A Web-based Intuitive Eating Intervention for Young Women With Disordered Eating: A Pilot Randomized Controlled Trial
Brief Title: Intuitive Eating for Disordered Eating
Acronym: IERCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeshiva University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20200516
Record Dates: First submitted 2021-07-14; First posted 2021-09-02 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Eating Disorder Symptom; Eating Behavior; Body Image; Psychological Distress
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intuitive Eating Treatment (Experimental): The intervention was a novel 10-week program aimed at promoting IE through pre-recorded videos, reading material, and bi-weekly discussion sessions. The intervention introduced the following modules sequentially: Unconditional Permission to Eat, Reliance to Hunger and Fullness Cues, Body-Food Choice Congruence, Gentle Nutrition, and Joyful Movement.
  Every other week, a new module was introduced. Participants were taught the concept of this module through video and reading, then prompted to practice it over the week. On opposite weeks, the module last introduced was discussed in greater detail through video, and participants were given the opportunity to discuss amongst one another and have all questions answered by the researchers.
  Interventions: Behavioral: Intuitive Eating Treatment
- Waitlist Control (No Intervention): Waitlist control group participants completed a series of questionnaires at the beginning and end of a 10-week interval, to compare changes in those who completed the intervention versus those who did not. This group was subsequently invited to participate in the intervention after their time on the wait-list.

INTERVENTIONS:
Behavioral: Intuitive Eating Treatment — Participants received a brief web-based intervention for disordered eating which focused on a style of eating behavior called "intuitive eating". Please see arm description for more details.
  Arms: Intuitive Eating Treatment

SUMMARY:
Purpose: Research on intuitive eating is growing, but there are few interventions demonstrating the effect of learning to eat intuitively for people with disordered eating. Young women in particular are at high-risk for developing disordered eating. This study aimed to test the outcomes of a novel intuitive eating intervention for young women with disordered eating.

Methods: This study is the first randomized controlled trial introducing intuitive eating to a sample of participants with disordered eating. Participants with current eating disorders were excluded from this study. Women (n=123) ages 18-30 with high levels of disordered eating participated in this study and were randomized to either a treatment (10-week web-based intervention) or control group (10-week waitlist).

ELIGIBILITY:
Inclusion Criteria:

* Female
* Between 18 and 30 years of age
* Located in the United States or Canada
* No eating disorder
* No previous participation in an intuitive eating intervention
* Score greater than or equal to 25 on the TFEQ-r18 at baseline

Exclusion Criteria:

* Gender not female
* Younger than 18 years of age
* Older than 30 years of age
* Located outside the United States or Canada
* Score less than 25 on the TFEQ-r18 at baseline
* Previously participated in an intuitive eating intervention
* Current eating disorder

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women are affected by disordered eating at higher rates than men.
Enrollment: 123 (Actual)
Dates: Start 2020-04-08 (Actual); Primary Completion 2020-09-02 (Actual); Study Completion 2021-03-17 (Actual)

PRIMARY OUTCOMES:
Intuitive Eating | Baseline (Time 1) through study completion, 10 weeks (Time 2)
  Intuitive eating was measured by the Intuitive Eating Scale, 2nd edition (IES-2). Scores on this scale range from 1 to 5, with higher scores indicating greater levels of Intuitive Eating.
Disordered Eating | Baseline (Time 1) through study completion, 10 weeks (Time 2)
  Revised Three Factor Eating Questionnaire (TFEQ-r18)

SECONDARY OUTCOMES:
Body Appreciation | Baseline (Time 1) through study completion, 10 weeks (Time 2)
  Body appreciation was measured by the Body Appreciation Scale, 2nd edition (BAS-2). Scores on this scale range from 13 to 65, with higher scores indicating greater levels of body appreciation.
Dichotomous Thinking Around Food | Baseline (Time 1) through study completion, 10 weeks (Time 2)
  Dichotomous thinking around food was measured by the Dichotomous Thinking Scale (DT). Scores on this scale range from 11 to 44, with higher scores indicating greater levels of dichotomous thinking around food.
Psychological Flexibility | Baseline (Time 1) through study completion, 10 weeks (Time 2)
  Psychological flexibility was measured by the Acceptance and Action Questionnaire, 2nd edition (AAQ-2). Scores on this scale range from 7 to 49, with higher scores indicating greater psychological flexibility.
Food Intake | Baseline (Time 1) through study completion, 10 weeks (Time 2)
  Food intake was measured by the NHANES Food Frequency Questionnaire (NHANES-FFQ), which collects data on respondents' food intake. Participants are asked to recall the frequency in which they consumed various food items over the past 3 days. Frequencies are grouped by food type (i.e., vegetables, fruits, dairy, etc.) and summed.
Body Mass Index (BMI) | Baseline (Time 1) through study completion, 10 weeks (Time 2)
  Weight/Height used to calculate BMI

CONTACTS AND LOCATIONS:
Locations (1):
- Study was conducted exclusively online, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available upon request to jduncan1@mail.yu.edu
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Researchers may request data after investigators publish results

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-15): https://cdn.clinicaltrials.gov/large-docs/11/NCT05031611/Prot_SAP_000.pdf
  • Informed Consent Form (2021-02-15): https://cdn.clinicaltrials.gov/large-docs/11/NCT05031611/ICF_001.pdf